CLINICAL TRIAL: NCT03742453
Title: Evaluation of Diagnostic Accuracy of Contrast-enhanced Ultrasound (CEUS) and Gadoxetic Acid-enhanced Liver MRI for Diagnosis of Hepatocellular Carcinoma in Patients With Liver Cirrhosis
Brief Title: Evaluation of Diagnostic Accuracy of CEUS for HCC Diagnosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Bracco Corporate (Industry)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SNUH-2018-2268
Record Dates: First submitted 2018-11-13; First posted 2018-11-15 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: CEUS; gadoxetic acid; MRI
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hepatic nodule group (Experimental): This group meets eligibility criteria, and undergo contrast-enhanced ultrasound (CEUS) and scheduled gadoxetic acid MRI (gadoxetic acid-enhanced liver MRI; EOB-MRI; Gd-EOB-MRI)
  Interventions: Diagnostic Test: contrast-enhanced ultrasound; Diagnostic Test: EOB-MRI

INTERVENTIONS:
Diagnostic Test: contrast-enhanced ultrasound — CEUS is performed using SonoVue (Bracco, Milan, Italy) intravenous administration in eligible participants within a month before/after EOB-MRI.
  Other Names: CEUS
Diagnostic Test: EOB-MRI — EOB-MRI is performed using standard dose of hepatocyte specific contrast media (primovist or eovist) according to standard protocol of our institution.
  Other Names: gadoxetic acid MRI; Gd-EOB-MRI

SUMMARY:
This study aims to compare the diagnostic accuracy of Contrast-enhanced ultrasound (CEUS) for diagnosing hepatocellular carcinoma (HCC) with that of gadoxetic acid-enhanced liver magnetic resonance imaging (MRI) using non-invasive diagnostic criteria (American Association for the Study of Liver Disease (AASLD or Liver Imaging Reporting and Data System (LI-RADS) v2018 and Korean Liver Cancer Study Group- National Cancer Center Korea (KLCSG-NCC) v2018).

ELIGIBILITY:
Inclusion Criteria:

* High risk group of developing HCC
* hepatic nodule equal to or larger than 1cm on ultrasound or computed tomography (CT)
* newly detected nodule (equal to or larger than 1cm, at least 2cm distance from radiofrequency ablation (RFA) site or resection margin) in patients with history of hepatic resection or RFA for HCC AND in remission more than a year
* scheduled for gadoxetic acid-enhanced liver MRI
* signed informed consent

Exclusion Criteria:

* hypersensitivity for ultrasound contrast media
* pregnancy
* history of recent treatment for HCC in a year
* standard of reference is not available
* severe cardiopulmonary disease (right to left shunt, severe pulmonary hypertension, uncontrolled hypertension, etc)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of CEUS for diagnosing HCC | 3 months after CEUS
  accuracy, sensitivity, specificity of CEUS for HCC diagnosis

SECONDARY OUTCOMES:
Diagnostic performance of gadoxetic-acid liver MRI for diagnosing HCC using LI-RADSv2018 | 3 months after MRI
  accuracy, sensitivity, specificity of MRI using LI-RADS v2018 for HCC diagnosis
Diagnostic performance of gadoxetic-acid liver MRI for diagnosing HCC using KLCSG-NCC guidelinev2018 | 3 months after MRI
  accuracy, sensitivity, specificity of MRI using KLCSG-NCC guideline v2018 for HCC diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No